CLINICAL TRIAL: NCT07259278
Title: Artificial Intelligence-enhanced Stratified Management Platform Guiding Home-based Exercise Rehabilitation for Coronary Heart Disease Patients: a Randomized Control Trial
Brief Title: Intelligent Management Platform for Guiding Exercise Rehabilitation in Coronary Heart Disease Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-I2M-C&T-B-040
Record Dates: First submitted 2025-11-14; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Secondary Prevention of Coronary Heart Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-Enabled Stratified Management Group (Experimental): Participants in the intervention group will receive comprehensive post-hospital rehabilitation management through an AI-based stratified management platform, utilizing a smartphone app and wearable device to track health data, deliver reminders and immediate safety alerts.
  Interventions: Combination Product: AI-Enabled Stratified Management System; Combination Product: Usual post-discharge care
- Standard Post-Discharge Care Group (Active Comparator): Participants in the control group will receive usual discharge protocol and personalized exercise prescription and goals from a specialist.
  Interventions: Combination Product: Usual post-discharge care

INTERVENTIONS:
Combination Product: AI-Enabled Stratified Management System — Following discharge, participants in the AI-stratified management group will use an intelligent platform (smartphone app + wearable divice) for home-based exercise rehabilitation and comprehensive post-discharge care. Key features include: 1) Safety Monitoring & Alerts: Real-time tracking of heart rate and other parameters via wristband triggers immediate safety warnings during exercise; 2) Holistic Risk Management: Integrated support for lifestyle modification, medication adherence, and control of cardiovascular risk factors; 3) Structured Engagement: Multi-channel reminders (messages, alarms, voice calls) for medications, exercise, and follow-ups to sustain adherence.
  Arms: AI-Enabled Stratified Management Group
Combination Product: Usual post-discharge care — Usual discharge protocol comprising verbal and printed discharge instructions addressing medication schedules, follow-up timelines, and lifestyle optimization strategies as well as a personalized exercise prescription.

SUMMARY:
The goal of this clinical trial is to find out if an artificial intelligence (AI)-enabled stratified management platform can help adults with coronary heart disease (CHD) better perform exercise rehabilitation and manage their health after being discharged from the hospital. The main questions it aims to answer are:

1. Does using the AI platform lead to a greater improvement in exercise capacity (measured by peak oxygen consumption, VO2peak) after 3 months?
2. Does the platform help increase daily physical activity, improve exercise adherence and motivation, and better control modifiable cardiovascular risk factors?
3. Is guiding home-based exercise with this platform safe for low-risk CHD patients?

Researchers will compare the AI Management Group (using the platform and a sports wristband) to the Routine Management Group (receiving usual care without the platform) to see if the AI group shows more significant improvements in fitness and health metrics.

Participants will:

1. Be randomly assigned to either use the AI platform or receive usual post-discharge care.
2. Receive a personalized exercise prescription from a doctor before going home.
3. If in the AI group: Use the smartphone app and wearable device to track health data for comprehensive post-discharge management, and receive reminders and immediate safety alerts.
4. Attend a follow-up visit at 3 months for check-ups and tests, including an exercise test and health assessments.

The study hopes to show that this intelligent management platform is an effective and safe tool to help people with CHD recover at home, stay active, and reduce future heart risks.

ELIGIBILITY:
Inclusion Criteria:

* CHD patients aged over 18 years;
* Stratified as low-risk for cardiovascular events during exercise and classified as low-risk according to the GRACE risk score.
* Ability of the patient or close relatives to use smartphones and applications;
* Willingness to participate and sign the informed consent form.

Exclusion Criteria:

* Residual stenosis of >50% in the left main coronary artery, or >70% stenosis in other major epicardial vessels;
* Planned coronary revascularization within the next 3 months;
* Acute myocardial infarction within the past 1 month;
* Severe cognitive impairment;
* Severely impaired exercise capacity.
* Advanced-stage malignancy;
* Life expectancy less than 3 months;
* Severe multi-organ failure;
* Other conditions deemed unsuitable for home-based exercise rehabilitation following assessment by a specialist rehabilitation physician.
* Refusal to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Peak oxygen consumption (VO2peak) | From enrollment to the end of treatment at 3 months.
  Peak oxygen consumption (VO2peak, mL∙kg-¹min-¹)

SECONDARY OUTCOMES:
Change in 6-minute walk distance | From enrollment to the end of treatment at 3 months
  6-minute walk distance (m)
Change in physical activity level (MET-min/week) | From enrollment to the end of treatment at 3 months
  Physical activity level (MET-min/week), estimated using the International Physical Activity Questionnaire-Short Form (IPAQ-SF). It consists of 7 questions with a recall period defined as 'last week'. The questions of the scale ask whether the participant walks for at least 10 minutes on any given day or does moderate or vigorous activities, and how much time/day the individual spends on each of these activities or sit.
Change in average daily step count | From enrollment to the end of treatment at 3 months
  Average daily step count (steps per day)
Exercise adherence | From enrollment to the end of treatment at 3 months.
  In the self-reported exercise diary, the participant will note the number of exercises done at home. The percentage adherence to the prescribed exercise regimen was calculated by dividing the number of exercises performed by the number of exercises prescribed and multiplying by 100.
Composite endpoints | From enrollment to the end of treatment at 3 months
  A composite endpoint including all-cause mortality, cardiac arrest, non-fatal myocardial infarction, and symptom-driven unplanned rehospitalization occurring during exercise. Safety endpoint during rehabilitation.
Systolic blood pressure (mmHg) | From enrollment to the end of treatment at 3 months
  Systolic blood pressure. Unit of Measure: mmHg.
Diastolic blood pressure (mmHg) | From enrollment to the end of treatment at 3 months
  Diastolic blood pressure. Unit of Measure: mmHg.
Glycated hemoglobin (HbA1c, %) | From enrollment to the end of treatment at 3 months
  Glycated hemoglobin. Unit of Measure: %.
Low-density lipoprotein cholesterol (LDL-C, mmol/L) | From enrollment to the end of treatment at 3 months
  Unit of Measure: mmol/L
Body mass index (BMI, kg/m^2) | From enrollment to the end of treatment at 3 months
Unplanned rehospitalization due to cardiovascular causes | From enrollment to the end of treatment at 3 months
Major Adverse Cardiovascular Events (MACE) | From enrollment to the end of treatment at 3 months
  Major Adverse Cardiovascular Events (MACE), defined as cardiovascular death, non-fatal myocardial infarction, and non-fatal stroke.
Anxiety level by Generalized Anxiety Disorder-7 scale score | From enrollment to the end of treatment at 3 months
  Anxiety level, assessed using the Generalized Anxiety Disorder-7 (GAD-7) questionnaire. Patients will be evaluated at the beginning and at the endpoint of the study with the self-administered GAD-7 scale. The GAD-7 scale score ranges from 0 to 21 points. A score between 5 and 9 points characterizes mild GAD. Between 10 and 14, moderate GAD and between 15 and 21, severe GAD.
Depression level by Patient Health Questionnaire-9 (PHQ-9) | From enrollment to the end of treatment at 3 months
  Depression level, assessed using the Patient Health Questionnaire-9 (PHQ-9). The GAD-7 scale score ranges from 0 to 27 points. A score between 5 and 9 points characterizes mild depression. Between 10 and 14, moderate depression; between 15 and 19, moderate-severe depression; and between 20 and 27, severe depression.
Sleep quality, assessed using the Pittsburgh Sleep Quality Index (PSQI) | From enrollment to the end of treatment at 3 months
  Sleep quality, assessed using the Pittsburgh Sleep Quality Index (PSQI). The total score ranges from 0 to 21 with a higher score indicating poor quality of sleep (worse). The higher the score, the worse the sleep quality. A cut-off score of >5 indicates poor sleep quality.
Quality of life by the EuroQol-5 Dimensions-5 Levels (EQ-5D-5L) questionnaire | From enrollment to the end of treatment at 3 months
  Quality of life, assessed using the EuroQol-5 Dimensions-5 Levels (EQ-5D-5L) questionnaire. This questionnaire asks 5 multiple-choice questions about mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. EQ-5D-5L index scores range from 0 to 100, where 100 is the best possible health state.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, Chinese Academy of Medical Sciences/National Center for Cardiovascular Diseases, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in publications will be shared, including all collected de-identified IPD.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available beginning 6 months after publication of the primary results and will remain available for at least 5 years thereafter.
Access Criteria: De-identified IPD and supporting documents will be made available upon reasonable request to the Principal Investigator (PI). Requests must include a methodologically sound proposal and intended use. Access will be granted at the discretion of the PI after review of the request.